CLINICAL TRIAL: NCT06186479
Title: Clinical Trial With Aconite Pain Oil in Oncology Patients Under Chemotherapy to Prevent Grade-II Chemotherapy-induced Polyneuropathy (CIPN), to Reduce Symptoms Typical of CIPN, and to Improve the Quality of Life of Patients With CIPN
Brief Title: Clinical Trial With Aconite Pain Oil in Oncology Patients Under Chemotherapy to Prevent CIPN Grade-II, to Reduce Symptoms and to Improve the Quality of Life of Patients With CIPN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: WALA Heilmittel GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: kp-acs-2
Record Dates: First submitted 2023-11-27; First posted 2024-01-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Chemotherapy-induced Polyneuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental)
  Interventions: Drug: Aconite pain oil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aconite pain oil — Participants apply 6 ml oil topically 2 times per day (morning and evening) for 15 to 27 weeks on chemotherapy-free days as long as they receive chemotherapy.
  Arms: Verum
Drug: Placebo — Participants apply 6 ml oil topically 2 times per day (morning and evening) for 15 to 27 weeks on chemotherapy-free days as long as they receive chemotherapy.
  Arms: Placebo

SUMMARY:
The clinical trial is planned as a prospective, multicentre, blinded, randomised, placebo-controlled, national clinical trial in Germany. The clinical trial is designed for testing the prophylactic and therapeutic effects of Aconite pain oil as compared to placebo in oncological patients receiving neurotoxic chemotherapy with taxanes and/or platinum derivatives.

ELIGIBILITY:
Inclusion Criteria:

1. A consent form, fully dated and signed by the patient and the principal investigator/investigator, is available
2. Patients with a minimum age of 18 years
3. Patients with a Karnofsky Index ≥ 70%
4. Patients with an assumed life expectancy of at least 12 months
5. Patients with solid tumours
6. Patients who are scheduled to receive unmodified chemotherapy with taxanes or platinum derivatives or their combination approved in Germany for at least 3 months (3 lunar months / 12 weeks)
7. Patients of childbearing age must provide a negative pregnancy test

Exclusion Criteria:

1. Participation in an interventional trial (with an investigational product) that is concurrent or occurred within 4 weeks prior to inclusion in this trial
2. Pregnant and breastfeeding patients or patients who are not using effective contraception (Pearl index < 1)
3. Patients treated with topical and/or internally administered medicinal products or cosmetics containing aconite (Aconitum napellus), camphor (Camphora), lavender essential oil (Lavandulae aetheroleum), and/or quartz within 4 weeks prior to inclusion in this trial
4. Patients with known hypersensitivity to camphor and/or any of the other ingredients of Aconite Pain Oil, as well as peanut or soy
5. Patients who are not expected to be able to comprehend the significance of the clinical trial, to demonstrate the necessary compliance, and/or to complete the patient questionnaire and patient diary in the German-language for language-related, cognitive, or other reasons
6. Patients with a planned application of chemotherapy at ≥4-week intervals
7. Patients with alcohol/drug/medication dependency
8. Patients with known genetic predispositions to polyneuropathies
9. Patients with previous or current polyneuropathy irrespective of cause
10. Patients with previous or current neurotoxic medication outside the planned chemotherapy protocol that has an impact on the primary endpoint (at the investigator´s discretion) and prior taxane and/or platinum derivative administration
11. Patients with the following known comorbidities that predispose them to CIPN:

    inadequately substituted hypothyroidism, renal insufficiency grade 4 and above, vasculitis/collagenosis, inadequately treated diabetes mellitus
12. Patients with active and/or clinically relevant infectious diseases: HIV, Lyme disease, hepatitis B/C, herpes infections
13. Known presence of multiple myeloma or non-Hodgkin's lymphoma
14. Present neurological diseases, Alzheimer's disease, multiple sclerosis, Parkinson's disease, and other neurological diseases that make it difficult or impossible to assess the primary endpoint according to the investigator's opinion
15. Patients with metastases in the central nervous system
16. History of amputation of extremities
17. Patients with distal muscle weakness and/or atrophy
18. Skin lesions or other findings in the area of the extremities that make it impossible to use the investigational product (e.g., hand-foot syndrome)
19. Presence of any other serious acute or chronic organic or mental illness with severe impairment of the general condition that impairs or prevents regular participation in the trial
20. Use of co-analgesics such as gabapentin, pregabalin, amitriptyline, nortriptyline, clomipramine, imipramine, duloxetine 1 week before commencement of the trial (baseline) and intake during the trial before reaching CIPN grade III
21. Planned acupuncture for the treatment of CIPN during the trial
22. Topical application of substances such as lidocaine, capsaicin, botulinum toxin, amitriptyline, menthol to hands and/or feet up to 1 week before trial entry (baseline) and application during the trial
23. Electrotherapy on the extremities up to 1 week before the start of the trial (baseline) and during the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of CIPN grade II and higher measured by "Common Terminology Criteria for Adverse Events" (CTC-AE v4.0 of 2010) | on average every 3 weeks for max. 27 weeks
  for neuralgia, paraesthesia, peripheral motor polyneuropathy, peripheral sensory polyneuropathy
The date of occurrence of CIPN by the principal investigator/investigator using the EORTC-QLQ-CIPN20 | on average every 3 weeks for max. 27 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medizinische Fakultät Mannheim der Uniklinik Heidelberg, Mannheim, Germany